CLINICAL TRIAL: NCT02065869
Title: Phase I/II Study of CaspaCIDe T Cells (BPX-501; Rivogenlecleucel) From an HLA Partially Matched Family Donor After Negative Selection of TCRαβ+ T Cells in Paediatric Patients Affected by Haematological Disorders
Brief Title: Safety Study of Gene Modified Donor T-cells Following TCRαβ+ Depleted Stem Cell Transplant
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Bellicum Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BP-004
Record Dates: First submitted 2014-02-13; First posted 2014-02-19 (Estimated); Results first posted 2023-01-04 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Acute Lymphoblastic Leukemia; Leukemia, Acute Myeloid (AML), Child; Lymphoma, Non-Hodgkin; Myelodysplastic Syndrome; Primary Immunodeficiency; Anemia, Aplastic; Osteopetrosis; Hemoglobinopathies; Cytopenia; Fanconi Anemia; Diamond Blackfan Anemia; Thalassemia; Anemia, Sickle Cell
Keywords: ALL; AML; hematologic neoplasms; hematologic malignancies; primary immune deficiences; hemoglobinopathy; congenital cytopenia; anemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia; Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin; Myelodysplastic Syndromes; Primary Immunodeficiency Diseases; Anemia, Aplastic; Osteopetrosis; Hemoglobinopathies; Cytopenia; Fanconi Anemia; Anemia, Diamond-Blackfan; Thalassemia; Anemia, Sickle Cell; Hematologic Neoplasms; Anemia | interventions — AP 1903 reagent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BPX-501 T cells and rimiducid (Experimental): TCR alpha beta depleted graft infusion with addback of BPX-501 T cells (rivogenlecleucel).
  Rimiducid/AP1903: Dimerizer drug administered to subjects who develop Grade III-IV acute GVHD, Grade II gut/liver acute GVDH or Grade I/II skin-only acute GvHD which is non-responsive after 7 days of standard of care treatment
  Interventions: Biological: BPX-501 T cells; Drug: Rimiducid

INTERVENTIONS:
Biological: BPX-501 T cells — 1x10E6 cells/kg infused on Day 0
  Other Names: Rivogenlecleucel
Drug: Rimiducid — 0.4mg/kg administered IV to treat GVHD
  Other Names: AP1903

SUMMARY:
This study will evaluate pediatric patients with malignant or non-malignant blood cell disorders who are having a blood stem cell transplant depleted of T cell receptor (TCR) alfa and beta cells that comes from a partially matched family donor. The study will assess whether immune cells, called T cells, from the family donor, that are specially grown in the laboratory and given back to the patient along with the stem cell transplant can help the immune system recover faster after transplant. As a safety measure these T cells have been programmed with a self-destruct switch so that they can be destroyed if they start to react against tissues (Graft versus host disease).

DETAILED DESCRIPTION:
This is a Phase I/II study evaluating the safety and feasibility of BPX-501 T cells infused after partially mismatched, related, TCR alpha beta T cell depleted hematopoietic stem cell transplant (HSCT) in pediatric patients. The purpose of this clinical trial is to determine whether BPX-501 infusion can enhance immune reconstitution in those patients with hematologic disorders, with the potential for reducing the severity and duration severe acute graft versus host disease (GvHD).

The trial will also evaluate the treatment of GvHD by the infusion of dimerizer drug (AP1903/rimiducid) in those subjects who present with GVHD who progress or do not respond to standard of care treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age < 18 years and > 1 month (< 1 month upon approval by Sponsor)
2. Life expectancy > 10 weeks
3. Patients deemed clinically eligible for allogeneic stem cell transplantation.
4. Patients may have failed prior allograft
5. Patients with life-threatening acute leukemia (high-risk ALL in 1st CR, ALL in 2nd CR, high-risk AML in 1st CR, AML in 2nd CR.) or myelodysplastic syndromes. Morphological CR must be documented and minimal residual disease measurement before transplantation is recommended.
6. Non-malignant disorders deemed curable by allogeneic transplantation: (a) primary immune deficiencies, (b) severe aplastic anemia not responding to immune suppressive therapy, (c) osteopetrosis, (d) selected cases of erythroid disorders such as β0 β0 thalassemia major, sickle cell disease, Diamond-Blackfan anemia, (e) congenital/hereditary cytopenia, including Fanconi Anemia before any clonal malignant evolution (MDS, AML).

   Note: Subjects will be eligible if they meet either item 5 OR item 6.
7. Lack of suitable conventional donor (HLA identical sibling or HLA phenotypically identical relative or 10/10 unrelated donor evaluated using high resolution molecular typing) or presence of rapidly progressive disease not permitting time to identify an unrelated donor
8. A minimum genotypic identical match of 5/10 is required.
9. The donor and recipient must be identical, as determined by high resolution typing, on at least one allele of each of the following genetic loci: HLA-A, HLA-B, HLA-Cw, HLA- DRB1 and HLA-DQB1.
10. Lansky/Karnofsky score > 50
11. Signed informed consent by the patient or the patient's parent or guardian for patients who are minors

Exclusion Criteria:

1. Greater than active Grade II acute GvHD or chronic extensive GvHD due to a previous allograft at the time of screening
2. Patient receiving an immunosuppressive treatment for GvHD treatment due to a previous allograft at the time of screening
3. Dysfunction of liver (ALT/AST > 5 times normal value, or bilirubin > 3 times normal value), or of renal function (creatinine clearance <30ml/min/1.73m2)
4. Severe cardiovascular disease (arrhythmias requiring chronic treatment, congestive heart failure or left ventricular ejection fraction < 40%)
5. Current clinically active infectious disease (including positive HIV serology or viral RNA)
6. Serious concurrent uncontrolled medical disorder
7. Pregnant or breast feeding female patient
8. Lack of parents'/guardian's informed consent for children who are minors.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 187 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2021-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bellicum Pharmaceuticals, Study Director — Bellicum Pharmaceuticals, Inc.
Locations (4):
- IRCCS Ospedale Pediatrico Bambino Gesù, Roma, Italy
- United Kingdom (3):
  - Royal Free London NHS Foundation Trust, London
  - Institute of Child Health & Great Ormond Street Hospital, London
  - Great North Children's Hospital, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- BPX-501 T Cells and Rimiducid: TCR alpha beta depleted graft infusion with addback of BPX-501 T cells (rivogenlecleucel).
  Rimiducid/AP1903: Dimerizer drug administered to subjects who develop Grade III-IV acute GVHD, Grade II gut/liver acute GVDH or Grade I/II skin-only acute GvHD which is non-responsive after 7 days of standard of care treatment
  BPX-501 T cells: 1x10E6 cells/kg infused on Day 0
  Rimiducid: 0.4mg/kg administered IV to treat GVHD
Period: Overall Study
Arm/Group | BPX-501 T Cells and Rimiducid
Started (Patients receiving HSCT graft (HSCT Safety population)) | 184
Patients Receiving Rivogenlecleucel (BPX-501 Safety Population) | 171
ITT Population | 142
Patients Receiving at Least 1 Dose of Rimiducid | 16
Completed | 149
Not Completed | 35
Not completed — Death | 7
Not completed — Disease relapse | 16
Not completed — Lost to Follow-up | 4
Not completed — No rivogenlecleucel cells infused (non-evaluable) | 7
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All enrolled patients iwho received HSCT (HSCT safety population)
Arm/Group | BPX-501 T Cells and Rimiducid
Number analyzed (Participants) | 184
Age, Continuous [Mean (Full Range); unit: years] — One patient was enrolled under a protocol version for which the inclusion criterion was <= 21 years and ≥ 3 months. The age range was revised in a subsequent protocol to < 18 years and ≥ 1 month (< 1 month upon approval by Sponsor).
  years | 5.8 [0.1 to 18.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83
  Male | 101
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 162
  More than one race | 1
  Unknown or Not Reported | 11

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS) at 180 Days After Transplant
Description: Events included transplant-related mortality (TRM) / non-relapse mortality (NRM), severe GvHD (acute Grades 2-4 organ or extensive chronic GvHD) and life-threatening infections (Grade 4). Time to the first event only is represented in the primary endpoint, if a subsequent event occurred in the same patient this was not captured in this outcome.
  There were no protocol-specified primary endpoints for Phase I of the study.
Time Frame: 180 days after transplant
Population: ITT population: All patients treated with HSCT who received 1×10^6 cells/kg BPX-501
Measure: Number (95% Confidence Interval); unit: Event-Free Survival Estimate (%)
Arm/Group | BPX-501 T Cells and Rimiducid
Number analyzed (Participants) | 142
Event-Free Survival Estimate (%) | 90.8 [84.6 to 94.5]

ADVERSE EVENTS:
Time Frame: Within 180 days post BPX-501 or 30 days post Rimiducid
Description: Analysis of All Cause Mortality was performed with the HSCT Safety Population (all patients who received a HSCT).
  Analysis of safety, regardless of study treatment and in relation to BPX-501, was conducted with the BPX-501 Safety Population (patients who received HSCT and subsequently received any dose of BPX-501) Analysis of safety in relation to rimiducid treatment was performed with the Rimiducid Population, (patients who received at least 1 dose of rimiducid)
Groups:
- BPX-501: BPX-501 (rivogenlecleucel): TCR alpha beta depleted graft infusion with addback of BPX-501 T cells
  BPX-501 T cells: 1x10E6 cells/kg infused on Day 0
- Rimiducid: Rimiducid/AP1903: Dimerizer drug administered to subjects who develop Grade III-IV acute GVHD, Grade II gut/liver acute GVDH or Grade I/II skin-only acute GvHD which is non-responsive after 7 days of standard of care treatment
  Rimiducid: 0.4mg/kg administered IV to treat GVHD
Arm/Group | BPX-501 | Rimiducid
All-Cause Mortality (participants affected / at risk) | 7/171 | 0/16
Serious Adverse Events (participants affected / at risk) | 52/171 | 7/16
Other Adverse Events (participants affected / at risk) | 140/171 | 9/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BPX-501 (N=171) | Rimiducid (N=16)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 2 | 0
Cytopenia (Blood and lymphatic system disorders) | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 2 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Pneumopericardium (Cardiac disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Parotid gland enlargement (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Device damage (General disorders) | 2 | 0
Malaise (General disorders) | 1 | 0
Medical device complication (General disorders) | 1 | 0
Pyrexia (General disorders) | 7 | 0
Acute graft versus host disease (Immune system disorders) | 4 | 2
Adenovirus infection (Infections and infestations) | 2 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 3 | 0
Device related infection (Infections and infestations) | 3 | 0
Encephalitis (Infections and infestations) | 2 | 0
Escherichia infection (Infections and infestations) | 2 | 0
Gastroenteritis rotavirus (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 1 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 2 | 0
Varicella zoster virus infection (Infections and infestations) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Juvenile chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Central nervous system lesion (Nervous system disorders) | 1 | 1
Encephalopathy (Nervous system disorders) | 1 | 1
Miller Fisher syndrome (Nervous system disorders) | 1 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cardiopulmonary failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 0
Pelvic venous thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BPX-501 (N=171) | Rimiducid (N=16)
Cytomegalovirus infection (Infections and infestations) | 34 | 0
Adenovirus infection (Infections and infestations) | 11 | 0
Human herpesvirus 6 infection (Infections and infestations) | 9 | 0
Acute graft versus host disease (Infections and infestations) | 48 | 3
Rash (Skin and subcutaneous tissue disorders) | 21 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 0
Diarrhoea (Gastrointestinal disorders) | 20 | 0
Vomiting (Gastrointestinal disorders) | 20 | 0
Nausea (Gastrointestinal disorders) | 10 | 0
Pyrexia (General disorders) | 33 | 0
Sepsis (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 1 | 1
Staphylococcal infection (Infections and infestations) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Parotid gland enlargement (Gastrointestinal disorders) | 1 | 1
Central nervous system lesion (Nervous system disorders) | 1 | 1
Encephalopathy (Nervous system disorders) | 1 | 1
Chronic graft versus host disease (Immune system disorders) | 5 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Right ventricular failure (Cardiac disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Confusional state (Psychiatric disorders) | 1 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-10-29): https://cdn.clinicaltrials.gov/large-docs/69/NCT02065869/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-08): https://cdn.clinicaltrials.gov/large-docs/69/NCT02065869/SAP_001.pdf